CLINICAL TRIAL: NCT06319833
Title: Effects of Brain Breaks on Educational Achievement in Children With and Without ADHD: The Break4Brain Project
Brief Title: Effects of Brain Breaks on Educational Achievement in School Settings: The Break4Brain Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); European Regional Development Fund (Other); State Research Agency, Spain (Other Government)
Responsible Party: Principal Investigator, Josep1, Senior Lecturer, University of the Balearic Islands
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 348CER23
Record Dates: First submitted 2024-02-02; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Physical Activity
Keywords: active breaks; executive functions; academic performance; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity interacting with a video (Experimental): This experimental condition involves engaging in physical activity interspersed with rest periods. The type of exercises are based on phase I.
  Interventions: Behavioral: Physical activity interacting with a video
- Control condition (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity interacting with a video — This experimental condition will be implemented five times a week, once per day, over 8 weeks. It will follow a structured format, including seven consecutive 40-second blocks of physical activity. The total video duration will amount to 9 minutes (40 seconds of activity followed by 20 seconds of rest, maintaining a 2:1 work-to-rest ratio). Additionally, participants will engage in 5 minutes of warm-up exercises and 5 minutes of cool-down activities. The experimental condition will consist of 10 videos, each centered around one of five different themes (a different one will be administered every day).
  Arms: Physical activity interacting with a video

SUMMARY:
A total of 600 children between 10 and 12 years of age will be randomized among two experimental conditions: physical activity interacting with a video (n = 300), and sedentary activity (n = 300). The experimental condition will take place in the school settings during the school day through a between-subject design with a total of two measurements, pre, and post-test. Using the latest advances, the transient effects of the experimental conditions on cognitive and academic performance will be measured. The experimental condition was crafted through a qualitative design involving semi-structured interviews with teachers (n = 41) and members of the management team (n = 16), along with questionnaires administered to students (n = 600). To enhance and ensure its sustainability, the same process will be replicated after the intervention. Interviews and questionnaires were meticulously crafted by the RE-AIM framework, and subsequently validated through a rigorous process involving an expert panel (n = 30) utilizing the Delphi methodology. This project has the potential to substantially contribute to the field of acute physical activity and could have a meaningful transference on the educational system. This method might be prescribed as an effective teaching strategy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-12 years.

Exclusion Criteria:

* Children who have serious physical or mental disorders (autism spectrum disorder, intellectual disability, and cerebral palsy) that would impede participation in the experimental conditions.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Academic achievement | 8 weeks
  Only the general academic fluency index was administered, consisting of the reading, mathematics, and writing fluency subtests. Reading fluency assessed the participant's capacity to read simple sentences rapidly, mathematical fluency gauged the ability to quickly solve simple addition, subtraction, and multiplication problems, and writing fluency measured the skill to formulate and write sentences promptly.
Inhibition-attention and cognitive flexibility | 8 weeks
  The assessment of inhibition-attention and cognitive flexibility was conducted using the "Trail Making Test".
Working memory | 8 weeks
  The measurement of working memory through "The Digit Memory Test," specifically focusing on auditory attention and verbal memory.
Selective attention | 8 weeks
  The measurement of selective attention within a limited timeframe was carried out using the "D2 test."
Design of active breaks: semi-structured questionnaires | 2 months (november and may)
  Pre- and post-intervention, to guarantee a proper design and future sustainability of the experimental condition, semi-structured questionnaires are administered to students. The responses are systematically categorized.
Design of active breaks: semi-structured interviews | 2 months (november and may)
  Pre- and post-intervention, to guarantee a proper design and future sustainability of the experimental condition, semi-structured interviews are administered to teachers and the management team. The responses are systematically categorized.

SECONDARY OUTCOMES:
Physical activity patterns | 8 weeks
  Physical activity patterns will be measured through accelerometry using the ActiGraph wGT3X-BT. Additionally, the intensity of the brain breaks will also be calculated with the same tool.
Self-report physical activity patterns | 8 weeks
  Physical activity levels over the preceding seven days were assessed using the PAQ-C.
Self-report sedentary patterns | 8 weeks
  Sedentary patterns over the preceding 7 days were assessed using the YAP-S.
Self-report physical fitness | 8 weeks
  The level of physical fitness was assessed using the self-administered IFIS questionnaire.
Socioeconomic level | 8 weeks
  The socioeconomic status was assessed through the Family Affluence Scale-II.
Student's behavior | 8 weeks
  The behavior of students in a regular classroom setting was examined using the "Child and Adolescent Behavior Inventory", inattention and hyperactivity-impulsivity parts, for teachers.
Body composition | 8 weeks
  Parents self-reported the body composition. In this case, parents will just report height (cm) and weight (kg).
Creativity | 8 weeks
  Participants were required to complete the maximum number of unusual uses for two objects within a 5-minute timeframe.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain